CLINICAL TRIAL: NCT03130478
Title: Predictors of Persistence in Patients With Schizophrenia Treated With Once-monthly Aripiprazole Long-acting Injection in the Spanish Clinical Practice: a Retrospective, Observational Study
Brief Title: Predictors of Persistence in Patients With Schizophrenia Treated With Once-monthly Aripiprazole in Spain
Acronym: PROSIGO
Status: Completed | Type: Observational
Sponsor: Otsuka Pharmaceutical Europe Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: 031-307-00162
Record Dates: First submitted 2017-04-21; First posted 2017-04-26 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Schizophrenia
Keywords: long-acting injectable antipsychotic; persistence
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

SUMMARY:
This is an observational, retrospective, non-interventional study that will include schizophrenic patients who were initiated on AOM treatment during an schizophrenia-related hospitalisation at least 6 months before data collection and in a real clinical practice setting.

DETAILED DESCRIPTION:
This is an observational, retrospective, non-interventional study that will include schizophrenic patients who were initiated on AOM treatment during an schizophrenia-related hospitalisation at least 6 months before data collection and in a real clinical practice setting.

Data from each patient will be collected after informed consent is obtained (if possible), and will include retrospective information mainly from the index date (start of AOM treatment, baseline timepoint) until the last information available in the patient file at the time of data collection (minimum of 6 months after the index date). Data will be retrospectively collected from all visits occurring as per clinical practice (usually once-monthly).

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (age ≥ 18 years at the time of AOM initiation).
2. Diagnosis of schizophrenia according to the Diagnostic and Statistical Manual of Mental Disorders V available at start of AOM treatment, and confirmed by the current investigator.
3. Having been hospitalized for an acute psychotic relapse and having been initiated with AOM as primary maintenance antipsychotic treatment, in accordance with the terms of the marketing authorisation, during the hospitalisation, at least 6 months before the inclusion and before November 1st 2016 (and up to January 2016 at the earliest).
4. Provision of patient informed consent unless a) not required by local regulations, b) it would take a non-reasonable effort* or c) if the source patient is deceased or untraceable.

   * A reasonable effort is defined as 3 contact attempts separated by 3 weeks. All efforts to obtain the informed consent, reasonable or not, shall be registered in the medical history of the patient to be used as documental source.

If allowable by Ethics Committees, provision of oral (e.g., by phone) instead of written consent is also possible for patients with retrospective assessment only.

Exclusion Criteria:

1. The patient has a psychiatric disorder other than schizophrenia which is established as the primary diagnosis
2. Chronically hospitalized patients at time of AOM initiation.
3. Patients who receive, after AOM initiation, a concomitant oral antipsychotic treatment for more than 4 weeks (with the exception of low dose quetiapine)*

   * Low dose quetiapine is acceptable up to a maximum of 150 mg daily only for sedative purposes, but not for the induction of any psychopharmacological effect on mood and/or psychosis.
4. Participation in an interventional clinical trial during the retrospective follow-up period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients will include adult patients with schizophrenia who have been initiated with AOM as primary maintenance AP treatment during an inpatient stay due to an acute schizophrenia relapse in a real clinical practice setting at least 6 months before the inclusion in the study (regardless of the current treatment at inclusion). Since persistence is part of the primary objective of the study, patients who discontinued the maintenance treatment with AOM before the inclusion period of the study should also be included.
Sampling Method: Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2017-07-18 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
Persistence (days) with aripiprazole once-monthly | First 6 months after treatment initiation
  To describe in real-world practice the impact of demographic and clinical characteristics on persistence in patients with schizophrenia initiated on aripiprazole once-monthly (AOM) during an inpatient stay due to an acute schizophrenia relapse.

SECONDARY OUTCOMES:
Description of reasons of treatment discontinuation (number of discontinuations per reason) | From treatment initiation up to patient inclusion (minimum 6 months)
  Date of AOM interruption or discontinuation and reason for discontinuation
Change over time in Clinical Global Impressions - Severity (CGI-S) scale | From treatment initiation up to patient inclusion (minimum 6 months)
  Clinical Global Impressions - Severity (CGI-S) scale at index date (if available in patient's file or estimated by the investigator according to medical records) and CGI-S up to patient's inclusion (if available in patients' file or estimated by the investigator according to medical records). CGI-S up to patient's inclusion (if available in patients' file or estimated by the investigator according to medical records).
Change over time in the Brief Psychiatric Rating Scale (BPRS) | From treatment initiation up to patient inclusion (minimum 6 months)
  Brief Psychiatric Rating Scale (BPRS) at index date (if available in patient's file) and BPRS up to the patient's inclusion (if available in patients' file).
Description of AOM treatment (starting dose and dose adjustments, number of injections, prior and concomitant medications, settings) | From treatment initiation up to patient inclusion (minimum 6 months)
  Description of AOM treatment (starting dose and dose adjustments, number of injections, prior and concomitant medications, settings)
Description of health resource use (HRU) related to schizophrenia (hospitalisations, medications, non-pharmacological therapies, outpatient visits, procedures) | From treatment initiation up to patient inclusion (minimum 6 months)
  Description of health resource use (HRU) related to schizophrenia (hospitalisations, medications, non-pharmacological therapies, outpatient visits, procedures)
Description of non-pharmacological interventions aiming to improve functionality (types, numbers of patients per type) | From treatment initiation up to patient inclusion (minimum 6 months)
  Description of non-pharmacological interventions aiming to improve functionality (including, if applicable, initiation and end dates of Institutional support, Cognitive behavioural therapy (CBT), Assertive Community Treatment/Case management, Group or individual psychoeducation, Family psychoeducation, Group or individual psychotherapy, Structured rehabilitation program, Occupational support, Severe mental illness management program)
Description of patterns of alcohol and drug abuse and/or dependence (patterns of drug abuse, type of substance, frequency of consumption) | From treatment initiation up to patient inclusion (minimum 6 months)
  To qualitatively describe patterns of drug abuse and/or dependence

CONTACTS AND LOCATIONS:
Overall Officials: Medical Department, Study Director — Otsuka Europe
Locations (15):
- Spain (15):
  - Hospital Universitario de Álava, Alava
  - Hospital Fundación Alcorcón, Alcorcón
  - Numància Salut Mental (Parc Sanitari St Joan de Deu), Barcelona
  - Hospital de Ciudad Real, Ciudad Real
  - Hospital IAS Girona, Girona
  - Hospital Universitari Bellvitge, L'Hospitalet de Llobregat
  - Complejo Asistencial Universitario de Leon, León
  - Fundación Jiménez Díaz, Madrid
  - HGU Gregorio Marañón, Madrid
  - Hospital Infanta Leonor, Madrid
  - Hospital Carlos Haya, Málaga
  - Parc Sanitari St. Joan de Deu (St. Boi), Sant Boi de Llobregat
  - Hospital Santiago de Compostela, Santiago de Compostela
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Álvaro Cunqueiro, Vigo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Olivares JM, Gonzalez-Pinto A, Paramo M; PROSIGO Study Group. Predictors of persistence in patients with schizophrenia treated with aripiprazole once-monthly long-acting injection in the Spanish clinical practice: a retrospective, observational study. Eur Psychiatry. 2021 Apr 12;64(1):e40. doi: 10.1192/j.eurpsy.2021.23. PMID 33840396